CLINICAL TRIAL: NCT04810676
Title: A Randomized, Open-label, Single-dose, Two-way Crossover Clinical Trial to Investigate the Pharmacokinetics and Safety After Oral Administration of CKD-383 and Co-administration of CKD-501, D745, D150 Under Fed Condition in Healthy Adults.
Brief Title: A Clinical Trial to Evaluate the Pharmacokinetic Profiles and Safety of CKD-383.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A101_02BE2020
Record Dates: First submitted 2021-03-11; First posted 2021-03-23 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Type2 Diabetes Mellitus
MeSH Terms: interventions — lobeglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): Peroid 1: CKD-501, D745, D150 -PO
  Peroid 2: CKD-383- PO
  Interventions: Drug: CKD-501, D745, D150; Drug: CKD-383
- Sequence 2 (Experimental): Peroid 1: CKD-383- PO
  Peroid 2: CKD-501, D745, D150 -PO
  Interventions: Drug: CKD-501, D745, D150; Drug: CKD-383

INTERVENTIONS:
Drug: CKD-501, D745, D150 — QD, PO
Drug: CKD-383 — QD, PO

SUMMARY:
A clinical trial to evaluate the pharmacokinetic profiles and safety of CKD-383.

DETAILED DESCRIPTION:
A phase 1 clinical trial to evaluate pharmacokinetics and safety in healthy adult after oral administration of CKD-383 and co-administration of CKD-501, D745, D150.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers aged between 19 and 55 years old.
2. Weight ≥ 55kg(men) or ≥50kg(women),
3. Calculated body mass index(BMI) of 18.5 to 27.0kg/m2

   * Body Mass Index(BMI) = Weight(kg) / [Height(m)]2
4. Women must meet one of the criteria written in below:

   * Menopause (No menstruation for 2 years)
   * Sterilization (hysterectomy or Oophorectomy, Tubal ligation etc.)
5. Men agree to contraception and not to donate sperm during the participation of clinical trial.
6. Those who voluntarily decide to participate and agree to comply with the cautions after fully understand of the detailed description of this clinical trial.

Exclusion Criteria:

1. Those who have a clinically significant disease or medical history of hepatic-biliary system issues, Renal dysfunction, Neurological disorder, Immunity disorder, Respiratory disorder, Genitourinary system disorder, Digestive system disorder, Endocrine system disorder, Cardiovascular disorder, Blood tumor and/or mental health problems.
2. Those who have signs and symptoms of clinically significant dehydration or who are vulnerable to dehydration by poor oral intake.
3. Those who receive intravenous administration of radioactive iodine contrast agents (for Urography, venous cholangiography, angiography, computed tomography using contrast agents, etc.) within 48hours before the first administration of investigational product.
4. Those who have severe urinary tract infection or have a past medical history of it.
5. Those who have genetic problems such as galactose intolerance, Lapp lactose deficiency or glucose-galactose malabsorption.
6. Those who have past medical history of gastrointestinal disorder(Crohn's disease, ulcerative colitis, etc. except simple appendectomy or hernia surgery), which affect the absorption of drug
7. Those who have history of hypersensitivity to active pharmaceutical ingredient(Lobeglitazone, Empagliflozin, Metformin) or additives.
8. Those who have the test results written in below:

   * AST/ALT > 1.25 times higher than upper normal level
   * eGFR(estimated Glomerular Filtration Rate, which is calculated by MDRD) < 60 mL/min/1.73m2
   * "positive" or "reactive" test result of Hepatitis B & C, HIV, PRP
   * Under 5 min resting condition, systolic blood pressure >150mmHg or <90mmHg, Diastolic blood pressure >100mmHg, or <50mmHg
9. Those who have a drug abuse history within one year or positive reaction on urine drug screening test
10. Those who received following drugs, which may affect results of clinical trial and safety. Ethical-the-counter (ETC) drugs and herbal medicines within 14 days before the first administration of the investigational drug. Over-the-counter (OTC) drugs, health foods and vitamin preparations within 7 days before the first administration of the investigational product.
11. Those who take barbiturate and related (causing induction or inhibition of metabolism) drug within 1 month before the first administration of investigational product
12. Those who exceeding an alcohol and smoke consumption criteria or can't stop smoking, consuming alcohol and caffeine during hospitalization period (Criteria: Caffeine > 5 cups/day, Alcohol > 210 g/week, Smoke > 10 cigarettes/day)
13. Those who took grapefruit before the first administration of investigational product or can't stop taking grapefruit during hospitalization period
14. Those who received investigational product by participating in other clinical trial within 6 months before the first administration of investigational product
15. Those who donated whole blood within 2 months or apheresis within 1 month
16. Those who received transfusion within 1 month
17. Those who are pregnant or breastfeeding
18. Those who are deemed inappropriate to participate in clinical trial by investigators

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
AUClast of CKD-383 | 0(pre-dose), 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 32, 48(hours)
  AUClast: Area under the concentration-time curve from time zero to the last measurable concetnration time
Cmax of CKD-383 | 0(pre-dose), 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 32, 48(hours)
  Cmax: Maximum plasma concentration of the drug

SECONDARY OUTCOMES:
AUCinf of CKD-383 | 0(pre-dose), 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 32, 48(hours)
  AUCinf: Area under the concentration-time curve from zero up to infinity
Tmax of CKD-383 | 0(pre-dose), 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 32, 48(hours)
  Tmax: Time to maximum plasma concentration
T1/2 of CKD-383 | 0(pre-dose), 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 32, 48(hours)
  T1/2: Terminal elimination half-life
Vd/F of CKD-383 | 0(pre-dose), 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 32, 48(hours)
  Vd/F: Volume of distribution
CL/F of CKD-383 | 0(pre-dose), 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 32, 48(hours)
  CL/F: Clearance

CONTACTS AND LOCATIONS:
Overall Officials: Min-soo Park, MD, PhD., Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, Yonsei-ro, Seodaemun-gu 50-1, South Korea